CLINICAL TRIAL: NCT00837148
Title: Phase II Trial of Sorafenib and Dacarbazine in Soft Tissue Sarcoma
Brief Title: Sorafenib and Dacarbazine in Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-068
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Sarcoma; Synovial Sarcoma; Leiomyosarcoma; Malignant Peripheral Nerve Sheath Tumor
Keywords: Sarcoma; Bone; BAY 43-9006 (SORAFENIB); DACARBAZINE; 08-068
MeSH Terms: conditions — Sarcoma; Sarcoma, Synovial; Leiomyosarcoma; Neurofibrosarcoma | interventions — Sorafenib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib and Dacarbazine (Experimental): This study is an open label, single arm, Simon two stage, phase 2 trial of continuous, daily oral sorafenib, with intravenous dacarbazine administered every three weeks for patients with synovial sarcoma, leiomyosarcoma and malignant peripheral nerve sheath tumor.
  Interventions: Drug: Sorafenib and Dacarbazine

INTERVENTIONS:
Drug: Sorafenib and Dacarbazine — Treatment will be administered on an outpatient basis. Sorafenib is supplied as 200-mg tablets. The starting dose of sorafenib will be 400 mg PO twice daily (every 12 hours) continuously. There is no planned treatment interruption between cycles.
  All patients will receive dacarbazine as an open-label dose of 850 mg/m2 by IV infusion over 60 minutes, starting on Week 1 and repeated every 3 weeks until disease progression or intolerance.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the combination of sorafenib and dacarbazine has on sarcoma. Recurrent sarcoma is difficult to treat. Standard chemotherapy drugs can be toxic, and the length of benefit is usually short. As a result, we need new treatments for sarcoma. Sorafenib is a new type of "targeted" chemotherapy that attacks specific proteins (including "raf" and "VEGF receptor") in cells. We hope that by blocking these proteins we can cause the tumor to shrink. Sorafenib is also known as BAY 43-9006 and by the trade name Nexavar®. The FDA approved sorafenib in December of 2005 to treat patients with kidney cancer and in November of 2007 to treat patients with liver cancer. This drug is not approved by the U.S. Food and Drug Administration (FDA) or any other licensing authority for the treatment of sarcoma and is therefore considered to be experimental in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed leiomyosarcoma, synovial sarcoma or malignant peripheral nerve sheath tumor (MPNST).
* Patients with metastatic, locally advanced, unresectable or locally recurrent disease.
* Zero to two prior chemotherapy regimens including neoadjuvant or adjuvant therapy.
* Measurable disease as defined by RECIST 1.1.
* Age ≥ 18.
* Karnofsky performance status of 50%-100%.
* Adequate bone marrow, liver and renal function as assessed by the following:

Hemoglobin ≥ 8.5 g/dl Absolute neutrophil count (ANC) ≥ 1,500/mm3 Platelet count ≥ 75,000/mm3 Total bilirubin < or = to 1.5 times ULN ALT and AST < or = to 2.5 times the ULN ( < or = to 5 x ULN for patients with liver involvement) Creatinine < or = to 1.5 times ULN

* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Patients should use adequate birth control for at least three months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* INR < 1.5 or a PT/PTT within normal limits if not on anticoagulation. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.

Exclusion Criteria:

* Prior therapy with dacarbazine, sorafenib or other antiangiogenic agents.
* Chemotherapy within 3 weeks or radiotherapy within 2 weeks of first day of protocol therapy.
* More than two prior chemotherapy regimens.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Pregnancy or nursing.
* Social situation or psychiatric illness that would limit compliance with study requirements.
* Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg for more than 24 hours, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection > CTCAE Grade 2.
* Thrombotic or embolic events such as a cerebrovascular accident, transient ischemic attack or myocardial infarction within the past 6 months, or deep venous thrombosis or pulmonary embolism within two months.
* Pulmonary hemorrhage/bleeding event > or = to CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > or = to CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any history of grade 4 thrombocytopenia (Plt <25,000), Grade 3 thrombocytopenia (Plt <50,000, >25,000) lasting 7 days or longer, or history of platelet transfusions for chemotherapy induced thrombocytopenia
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow pills.
* Any malabsorption problem that in the opinion of the investigator would interfere with the patients ability to tolerate oral sorafenib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tap, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Soft Tissue Sarcoma Patients: Sorafenib and Dacarbazine in Soft Tissue Sarcoma
Period: Overall Study
Arm/Group | Soft Tissue Sarcoma Patients
Started | 37
Completed | 35
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Soft Tissue Sarcoma Patients
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
Time Frame: at 18 weeks
Measure: Number; unit: participants
Arm/Group | Soft Tissue Sarcoma Patients
Number analyzed (Participants) | 35
participants
  Partial Response (PR) | 5
  Stable Disease (SD) | 22
  Progression of Disease (POD) | 8

ADVERSE EVENTS:
Arm/Group | Soft Tissue Sarcoma Patients
Serious Adverse Events (participants affected / at risk) | 8/37
Other Adverse Events (participants affected / at risk) | 30/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soft Tissue Sarcoma Patients (N=37)
Death not associated w CTCAE term- Death NOS (General disorders) | 1 (1)
Death not associated w CTCAE term-Disease progression NOS (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 2 (3)
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 1 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (2)
Obstruction of airway-Bronchus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain - Extremity-limb (General disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 2 (3)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soft Tissue Sarcoma Patients (N=37)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (3)
Amylase (Metabolism and nutrition disorders) | 3 (3)
Creatinine (Metabolism and nutrition disorders) | 3 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 7 (7)
Hemoglobin (Blood and lymphatic system disorders) | 10 (10)
Hypertension (Cardiac disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 19 (19)
Lymphopenia (Blood and lymphatic system disorders) | 14 (14)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 20 (20)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 15 (15)
Platelets (Blood and lymphatic system disorders) | 12 (12)
Potassium, low (hypokalemia) (Investigations) | 2 (2)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 7 (8)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes